CLINICAL TRIAL: NCT07289763
Title: Phase II Randomized, Open-label, Multicenter Clinical Study Evaluating the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of SHR-2173 Injection in Patients With Primary Membranous Nephropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-2173-201
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Primary Membranous Nephropathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-2173 injection
- Treatment group B (Experimental)
  Interventions: Drug: SHR-2173 injection
- Treatment group C (Experimental)
  Interventions: Drug: SHR-2173 injection

INTERVENTIONS:
Drug: SHR-2173 injection — SHR-2173 injection, with a total of 8 administrations
  Arms: Treatment group A
Drug: SHR-2173 injection — SHR-2173 injection, with a total of 16 administrations
  Arms: Treatment group B
Drug: SHR-2173 injection — SHR-2173 injection , with a total of 32 administrations
  Arms: Treatment group C

SUMMARY:
To investigate the safety, efficacy, pharmacokinetics, and pharmacodynamics of SHR-2173 injection in patients with primary membranous nephropathy

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, regardless of gender;
2. Weight ≥40.0 kg at screening;
3. Diagnosed as primary membranous nephropathy through kidney biopsy.

Exclusion Criteria:

1. Secondary membranous nephropathy.
2. Subjects developed rapidly progressive glomerulonephritis or required kidney transplantation.
3. Subjects who have undergone kidney dialysis in the previous 12 months or are expected to require dialysis during the study period.
4. Subjects who have a malignant tumor or a history of malignant tumor
5. Subjects who have undergone major surgery within the previous 3 months, or plan to undergo major surgery during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Week0, 2, 4, 8, 12,16, 20, 24, 28, 32, 36, 40, 48 52
12-lead ECG | Week4, 8, 12, 24, 28, 36, 52

SECONDARY OUTCOMES:
The proportion of subjects who achieved overall response (including complete response (CR) and partial response (PR)). | Week 12, 24, 36, 52
The proportion of subjects who achieved CR | Week 12, 24, 36, 52
The proportion of subjects who achieved PR | Week 12, 24, 36, 52

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital of eastern theater command, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided